CLINICAL TRIAL: NCT00710281
Title: Hemodynamic Analysis Of Intracranial Artery And Associated Lesions Using 2-D/3D Phase Contrast MR Angiography Focused On Wall Shear Stress Measurement
Brief Title: Analysis Of Intracranial Artery Lesions Using 2-D/3D Phase Contrast MR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator is no longer at study site
Sponsor: Lahey Clinic (Other)
Collaborators: VasSol®-Nova Software (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-020
Record Dates: First submitted 2008-07-01; First posted 2008-07-04 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Intracranial Arterial Aneurysm
Keywords: Intracranial Aneurysm; Subarachnoid arterial aneurysm; Aneurysm; Brain Aneurysm; Cerebral Aneurysm; Wall Shear Stress(WSS); Hemodynamic Stress; Subarachnoid Hemorrhage(SAH)
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2D/3D Phase contrast MR (Other)
  Interventions: Radiation: Additional scan time on standard MR angiography

INTERVENTIONS:
Radiation: Additional scan time on standard MR angiography — Procedure/Surgery: Additional 5 minutes scan time to standard MR angiography
  Using the Nova® Software, an additional 5 minutes scan time will be required in order to identify aneurysm, select target artery, and complete measurements
  Arms:
  Other Names: MRI; Phase contrast MR; 2D MR; 3D MR

SUMMARY:
Using phase contrast MR Angiography with NOVA® Software, this study intends to identify,evaluate and map intracranial aneurysm development as well as develope a predicator for future morphological changes of aneurysms and possible risk of future rupture.

DETAILED DESCRIPTION:
Hemodynamic stress toward the wall of intracranial artery with associated genuine defects of wall remodeling capacity is one of many hypotheses of subarachnoid aneurysm development. In addition, hemodynamic stress toward an aneurysm wall may play a very significant role for the rupture of an aneurysm creating acute Subarachnoid hemorrhage. We think the Wall Shear Stress (WSS) measurement toward an intracranial arterial wall and intracranial aneurysmal wall may provide valuable information for understanding of intracranial aneurysm development as well as predicting future morphological changes of aneurysm and possibly risk of future rupture. This study is significant especially in the management of unruptured subarachnoid arterial aneurysm patients and identifying patients who have higher rupture risks for active treatments such as surgical clipping or coiling to prevent unnecessary but potentially risky procedures.

Gadolinium MR Angiography with NOVA® Software will be used to measure the arterial wall shear stress (WSS) for patients with an intracranial arterial aneurysm. The aneurysm will be identified, blood flow, velocity, volume, vascular diameter and the direction of blood measurements will be taken using NOVA® Software at each point of interest. A WSS map of target intracranial artery and/or aneurysm sac will be created and matched with morphological features providing a clue to understand the the relationships between hemodynamic parameters, especially WSS and morphological changes.

ELIGIBILITY:
Inclusion Criteria:

* Unruptured and ruptured adult (>18 years) intracranial arterial aneurysm patients

Exclusion Criteria:

* Less than 18 years old
* Chronic renal failure patients
* Incompetent patient who cannot give consent for routine phase contrast MR Angiography and his/her surrogate decision maker is not available
* Any patients with a contraindication to having a standard MRI examination, such as phase maker, orbital metallic foreign body, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Identify, measure and map the Wall Shear Stress (WSS) measurements and affects in subarachnoid aneurysm developement. | Duration of the MRA test

SECONDARY OUTCOMES:
Develope predictor to identify risk factors of possible future aneurysm rupture and SAH | Duration of MRA test

CONTACTS AND LOCATIONS:
Overall Officials: Seon Kyu Lee, M.D., Ph.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Amin-Hanjani S, Du X, Zhao M, Walsh K, Malisch TW, Charbel FT. Use of quantitative magnetic resonance angiography to stratify stroke risk in symptomatic vertebrobasilar disease. Stroke. 2005 Jun;36(6):1140-5. doi: 10.1161/01.STR.0000166195.63276.7c. Epub 2005 May 12. PMID 15890993
- [Background] Zhao M, Amin-Hanjani S, Ruland S, Curcio AP, Ostergren L, Charbel FT. Regional cerebral blood flow using quantitative MR angiography. AJNR Am J Neuroradiol. 2007 Sep;28(8):1470-3. doi: 10.3174/ajnr.A0582. PMID 17846193
- [Background] Ahn S, Shin D, Tateshima S, Tanishita K, Vinuela F, Sinha S. Fluid-induced wall shear stress in anthropomorphic brain aneurysm models: MR phase-contrast study at 3 T. J Magn Reson Imaging. 2007 Jun;25(6):1120-30. doi: 10.1002/jmri.20928. PMID 17520716